CLINICAL TRIAL: NCT05975307
Title: A Single-arm, Phase II Clinical Trial to Treat Muscle-invasive Bladder Cancer With Neoadjuvant Chemotherapy Plus Anti-PD-1 Therapy Followed by Radiotherapy Plus Concurrent Anti-PD-1 Therapy
Brief Title: Treating Muscle-invasive Bladder Cancer With A Non-surgical Method Consisting of Anti-PD-1 Therapy and Chemoradiation
Acronym: BCIRT-01
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Vice Director of the Department of Radiation Oncology, Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-068
Record Dates: First submitted 2023-07-27; First posted 2023-08-03 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Programmed Cell Death Protein 1 Inhibitor; Radiotherapy
Keywords: Bladder Cancer; Programmed Cell Death Protein 1 Inhibitor; Radiotherapy; Chemotherapy; Bladder Preservation
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — toripalimab; Gemcitabine; Cisplatin; Carboplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: This phase 2 trial is an open-label, single-arm, non-comparative trial, in which all eligible patients will receive neoadjuvant chemotherapy plus toripalimab, followed by radiotherapy plus concurrent toripalimab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus chemoradiation (Experimental): This study has only single arm in which the patients will receive neoadjuvant chemotherapy plus anti-PD-1 therapy (toripalimab), followed by radiotherapy plus concurrent anti-PD-1 therapy
  Interventions: Drug: Toripalimab; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin; Radiation: Intensity-modulated radiation therapy

INTERVENTIONS:
Drug: Toripalimab — The patients in this arm will receive 3 cycles of neoadjuvant treatment containing chemotherapy with gemcitabine and cisplatin/carboplatin, plus toripalimab. Then the ones without progressive disease will receive radical radiotherapy, plus 2 cycles of concurrent toripalimab.
  Toripalimab: 240 mg on Day 1, every 3 weeks, totally 3 and 2 cycles in the neoadjuvant and concurrent phases, respectively.
  Other Names: JS001
Drug: Gemcitabine — The patients in this arm will receive 3 cycles of neoadjuvant treatment containing chemotherapy with gemcitabine and cisplatin/carboplatin, plus toripalimab. Then the ones without progressive disease will receive radical radiotherapy, plus 2 cycles of concurrent toripalimab.
  Gemcitabine: 1 g/m2 on Days 1 and 8, repeated every 3 weeks, totally 3 cycles.
Drug: Cisplatin — The patients in this arm will receive 3 cycles of neoadjuvant treatment containing chemotherapy with gemcitabine and cisplatin/carboplatin, plus toripalimab. Then the ones without progressive disease will receive radical radiotherapy, plus 2 cycles of concurrent toripalimab.
  Cisplatin: Used when creatinine clearance rate ≥ 40 ml/min, 37.5 mg/m2 on Days 1 and 2, repeated every 3 weeks, totally 3 cycles.
Drug: Carboplatin — The patients in this arm will receive 3 cycles of induction treatment containing chemotherapy with gemcitabine and cisplatin/carboplatin, plus toripalimab. Then the ones without progressive disease will receive radical radiotherapy, plus 2 cycles of concurrent toripalimab.
  Cisplatin: Used when creatinine clearance rate < 40 ml/min, area under curve = 2 on Days 1 and 2, repeated every 3 weeks, totally 3 cycles.
Radiation: Intensity-modulated radiation therapy — The patients in this arm will receive 3 cycles of neoadjuvant treatment containing chemotherapy with gemcitabine and cisplatin/carboplatin, plus toripalimab. Then the ones without progressive disease will receive radical radiotherapy, plus 2 cycles of concurrent toripalimab.
  Radiotherapy: performed by using the technique of intensity-modulated radiation therapy, with a total dose of 65 and 45 Gy for the gross tumor and lymphatic drainage regions.

SUMMARY:
The goal of this Phase 2 trial is to evaluate a non-surgical bladder-preserving treatment mode which consists of neoadjuvant chemotherapy plus anti-programmed cell death protein 1 (anti-PD-1) therapy followed by radiotherapy plus concurrent anti-PD-1 therapy. The main questions it aims to answer are: (i) whether the anti-PD-1 antibody, toripalimab, is effective in treating muscle-invasive bladder cancer (MIBC), when combined with chemoradiation; (ii) whether toripalimab is safe in combination with chemoradiation. Participants will receive 3 cycles of neoadjuvant treatment containing chemotherapy with gemcitabine and cisplatin/carboplatin, plus toripalimab. Then the ones without progressive disease will receive radical radiotherapy plus 2 cycles of concurrent toripalimab.

DETAILED DESCRIPTION:
Bladder cancer is the second most common malignancies over the world. At initial diagnosis, the cases with muscle-invasive bladder cancer (MIBC) accounts nearly 20% of all bladder cancer patients. And 40% of non-muscle-invasive bladder cancer could develop to MIBC. Currently, radical cystectomy (RC) is the golden standard to manage MIBC. Yet, it brings severe surgical injuries and post-surgical complications which impair life quality of the patients. Recently, bladder-preserving treatment based gradually becomes the second choice for MIBC. It consists of maximal transurethral resection of bladder tumor (TURBT) and chemoradiation. A series of clinical trials and meta-analyses supported that the bladder-preserving treatment has a similar therapeutic effect compared with RC. But it is noteworthy that this treatment mode does not really avoid surgery. TURBT could also cause complications, such as haemorrhage, infection, perforation, and even tumor dissemination. Moreover, the incidence of serious toxicities brought by concurrent chemoradiation is as high as 36%. In actual clinical work, it is hard for more than half patients to complete chemoradiation of standard intensity. Additionally, many patients are unsuitable for bladder preservation, including those with T stage > T2, diameter > 5 cm, hydronephrosis and positive lymph nodes. Hence, it calls for improvement of current bladder preservation mode, to make more MIBC patients receive radical treatment which brings better therapeutic experience and life quality.

Many lab studies indicated that formation and progression of bladder cancer is a process of mutation accumulation. It provides biological fundamentals for immune checkpoint inhibitors, such as anti-programmed cell death protein 1 (anti-PD-1) antibodies. Based on available clinical studies, anti-PD-1 antibodies exhibits ideal therapeutic effects in bladder cancer of different stages and has an incidence of toxicities as low as 13%. Its toxicities mainly include arthralgia and hyponatremia, which are well tolerated. Currently, there are more than 10 clinical trials trying anti-PD-1 antibodies for bladder preservation. However, the treatment modes in most of them still contain TURBT. This phase 2 trial intended to evaluate the therapeutic and adverse effects of a non-surgical bladder-preserving treatment mode consisting of anti-PD-1 antibodies and chemoradiation, in a small patient cohort with MIBC. The results might provide an effective, non-invasive and low-toxic choice which improves patient experience and realizes bladder preservation.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed bladder malignant tumor via biopsy
* Urothelial carcinoma as the primary histological component
* Pretreatment clinical TNM stage as T2-4aN0M0 or T1-4aN1-2M0 (UICC TNM staging classification, version 8)
* Age between 18 and 75 years old
* Karnofsky performance score ≥ 70
* Creatinine clearance rate ≥ 30 ml/min

Exclusion Criteria:

* Simultaneous tumors of the urethra or upper urinary tract
* Existence of small cell cancer component
* Uncontrolled tuberculosis, viral hepatitis or AIDS
* Autoimmune or mental diseases
* Severe cardiac, renal, hepatic or hematopoietic dysfunctions unsuitable for chemotherapy, radiotherapy or immune checkpoint inhibiting therapy
* Prior history of other malignancies within 5 years, except cured cervical carcinoma in situ and skin basal cell carcinoma
* Prior history of pelvic radiotherapy or chemotherapy
* Poor adherence to regular follow-up (cystoscopy, CT, MRI, etc.)
* Pregnant or lactating women
* Treatment with glucocorticoid or immunosuppressive drugs within 1 month
* Other situations for which the investigators consider a patient inappropriate to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical complete response (cCR) rate | When the eligible patients complete the treatment and followed-up for half a year
  The percentage of the cases attaining cCR of primary tumor and regional lymph nodes (confirmed by radiologic examinations, such as thoraco-bdominal computed tomography, pelvic magnetic resonance imaging, and multipoint biopsy under cystoscopy)

SECONDARY OUTCOMES:
Overall survival (OS) | When the eligible patients complete the treatment and followed-up for 1 and 2 years
  The percentage of the cases surviving over a given time period
Bladder-intact event-free survival (BI-EFS) | When the eligible patients complete the treatment and followed-up for 1 and 2 years
  The percentage of the cases surviving with intact bladder and without muscle-invasive recurrence, regional lymph node recurrence or distant metastasis, over a given time period
Disease-free survival (DFS) | When the eligible patients complete the treatment and followed-up for 1 and 2 years
  The percentage of the cases surviving without locoregional recurrence or distant metastasis over a given time period
Local recurrence (LR) rate | When the eligible patients complete the treatment and followed-up for 1 and 2 years
  The percentage of the cases with locoregional recurrence over a given time period
Incidence of grade 3/4 (G3/4) toxicities | Once a week during treatment, and once per 3 months after treatment, until the last follow-up (2 years after treatment)
  The percentage of the cases with any G3/4 toxicity during and after treatment
Bladder function | Once per 3 months after treatment, until the last follow-up (2 years after treatment)
  The quantitative score of bladder function at a given time point, based on the Quality of Life 30-item Questionnaire, Bladder Module (QLQ-BLM30) from the EORTC
Objective response rate (ORR) | A week before radiotherapy, and once per 3 months after treatment, until the last follow-up (2 years after treatment)
  The percentage of the cases attaining clinical complete or partial response of primary tumor and regional lymph nodes (confirmed by radiography and cystoscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Yuanhong Gao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China